CLINICAL TRIAL: NCT06131151
Title: Comparison Between Analgesic Effect of Ultrasound Guided External Oblique Intercostal Block and Erector Spinae Plane Block in Patients Undergoing Percutaneous Nephrolithotomy.
Brief Title: Comparison Between External Oblique Intercostal Block and Erector Spinae Plane Block in PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Gomaa Ismail, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EOI Block
Record Dates: First submitted 2023-10-30; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Oblique Intercostal Block (Experimental): 27 patients will receive External Oblique Intercostal Block. A volume of 20 ml of LA (20 ml of bupivacaine 0.375% plus 5 ug/ml adrenaline ) will be injected.
  Interventions: Other: Nerve block
- Erector Spinae Plane Block (Experimental): 27 patients will receive Erector Spinae Plane Block. A volume of 20 ml of LA (20 ml of bupivacaine 0.375% plus 5 ug/ml adrenaline ) will be injected.
  Interventions: Other: Nerve block

INTERVENTIONS:
Other: Nerve block — Nerve block in percutaneous nephrolithotomy

SUMMARY:
The aim of the study is to compare the post-operative analgesic effect of USG unilateral External oblique intercostal (EOI) block with Erector spinae plane block (ESPB) for after percutaneous Nephrolithotomy with a hypothesis that both External oblique intercostal fascial plane block and Erector spinae plane block are effective in providing postoperative analgesia.

DETAILED DESCRIPTION:
Introduction:

Percautaneous nephrolithotomy is the tretment of choice for patients with multiple or complex kidney or upper urinary tract stones. visceral pain from the kidney and ureter and somatic pain from the incision site are the primary cause of immediate postoperative pain following PCNL. poor pain control is associated with unwanted consequences such as patient discomfort, delayed recovery, and prolonged hospital stay.

This necessitates meticulous multi-modality analgesia due to mild to moderate pain originating from renal capsule dilatation or nephrostomy tube-related stress during the first 24 h after operation. Multimodal analgesia techniques are utilized broadly to manage postoperative pain. The concept of multimodal analgesia implies not only providing analgesic drugs, but also performing nerve blocks with local anaesthetics.

first described the Erector Spinae Plane Block (ESPB), the indications and clinical use of the block for different surgical interventions have been growing. Although ESPB is interfacial plane block, anatomical studies support the idea that some of its clinical benefit may derive from spread to the paravertebral and epidural space. External oblique intercostal (EOI) block is relatively new block technique modified aiming at obtaining upper midline and lateral abdominal wall analgesia. EOI block is achived by injecting the local anesthetic solution into the fascial plane on the deep aspect of the external oblique muscle. Previous studies have hypothesized that the block succesfully anesthetized the lateral cutaneous branch and the anterior cutaneous branch of the thoracoabdominal nerves, with low pain scores and minimal narcotic use postoperatively.

Recently, there have been several publications describing external oblique nerve blocks to control post-operativte pain after abdominal surgery.

Aim of the work:

The aim of this study is to compare the post-operative analgesic effect of USG unilateral External oblique intercostal (EOI) block with Erector spinae plane block (ESPB) for after Percutaneous Nephrolithotomy with a hypothesis that both External oblique intercostal fascial plane block and Erector spinae plane block are effective in providing postoperative analgesia.

Sample size calculation:

Based on the results of a previous study, a sample size of 21 patients in each group will be calculated to detect a 20% difference in the time to first analgesic request, with alfa=0.05 and a power of 85%. Twenty-seven patients in each group will be recruited to compensate for the dropouts.

Group A: will include 27 patients, will receive External Oblique Intercostal Block.

Group B: will include 27 patients, will receive Erector Spinae Plane Block. Randomization will be performed using an online random number generator. concealment was achieved using sealed opaque envelopes.

A) Anesthesia induction:

Standard monitoring procedures will include pulse oximetry, electrocardiography, and noninvasive arterial pressure prior to anesthetic induction. All patients will be premedicated with intravenous (i.v.) midazolam 1-2 mg and antibiotic prophylaxis, according to the hospitals protocol. Anesthesia will be induced with intravenously (IV) adminestrated propofol. 2mg/kg, fentanyl 1mic/kg, and recuronium bromide 0.6 mg/kg following which endotracheal intubation will be performed. Anesthesia will be maintained with oxygen, air, and isoflurane using controlled ventilation with closed circuit in order to ensure normocarbia. At the end of the surgery, patients will receive their intervention according to gorup allocation under sterile conditions.

B) Intervention:

1. External Oblique Intercistal Block:

   A high frequency linear ultrasound probe will be placed in a longitudinal parasagital orientation in the anterior midaxillary line. A 21G 10 cm needle will be inserted using an in-plane approach. The tip of the needle will be placed into the fascial plane on the deep aspect of the external oblique muscle. A volume of 20 ml of LA (20 ml of bupivacaine 0.375% plus 5 ug/ml adrenaline. ) will be injected.
2. Erector Spinae Plane block:

A high frequency linear ultrasound probe will be placed in a longitudinal parasagital orientation 2.5-3 cm lateral to the T9 spinous process. A 21G 10 cm needle will be inserted using an in-place approach. The tip of the needle will be placed into the fascial plane on the top of the aspect of the erector spinae muscle. A volume of 20 ml of LA (20 ml of bupivacaine 0.375% plus 5 ug/ml adrenaline. ) will be injected.

Peimary Outcome:

The first call for rescue analgesia.

Secondary Outcome:

1. The total analgesic requirement in 24 hours.
2. Any adverse effects related to anesthesia or the technique.
3. Pain scores; Numerical Rating Scales (NRS) at rest and when coughing (at 1, 2, 4, 8, 16 and 24 hours postoperatively.)
4. Block related complications during and after block procedure till 24 hours postoperatively (local anesthetic systemic toxicity, pneumothorax and vascular puncture during block procedure).

Statistical Analysis:

Continous data with normal distribution will be compared by paired or unpaired t-tests, whereas non-normally distributed data will be assessed using the Mann- Whitney U test and Wilcoxon ranksum test for unpaired and paired results, respectively. Chi-square test or fisher's exact test will measure the association between qualitative variables.

P-valve>0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years Body mass index of 18-35 kg/m2 Patients with the American Society of Anesthesiologists physical status I/II Patients scheduled for elective Percutaneous Nephrolithotomy Both sexes, males and females

Exclusion Criteria:

* Patients refusal Allergy to local anaesthetics Infection at the site of injection Coagulopathy Chronic pain syndrome Prolonged opioid medication Patients who received any analgesic 24 h befor surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The first call for rescue analgesia after the end of the surgery | 24 hours

SECONDARY OUTCOMES:
pain scores; Numerical Rating Scale (NRS) | 24 hours
  Numerical Rating Scale at rest and when coughing

CONTACTS AND LOCATIONS:
Overall Officials: Amr Thabet, Study Director — Department of anesthesia, intensive care and pain management